CLINICAL TRIAL: NCT03964571
Title: Human and Bacterial Protease Activity As Prognostic Tool of Foot Infections in Diabetic Patients
Acronym: CHEK BAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI GCS MERRI/2017/CDR-01
Record Dates: First submitted 2019-05-24; First posted 2019-05-28 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Foot Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diabetic foot patients (Experimental)
  Interventions: Diagnostic Test: WOUNDCHEK

INTERVENTIONS:
Diagnostic Test: WOUNDCHEK — fluid swab of wound and measurement of wound onto film

SUMMARY:
This study will establish whether human and bacterial protease activity can aid therapeutic decision-making, including targeted treatments.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient has been informed about the study objectives and purpose and their rights as a patient
* The patient is being treated in the Diabetes and Infectious Disease Department
* The patient has a chronic foot and/or heel wound classified as Grade 1-3 according to the Infectious Diseases Society of America.

Exclusion Criteria:

* The subject is participating in another category I interventional study, or has participated in another category I interventional trial in the previous 3 months, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant or breastfeeding
* The patient has chronic foot and/or heel wound classified as Grade 4 according to the Infectious Diseases Society of America
* Patient with critical ischemia defined by PSGo <50 mmHg or PSCh <70 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Reduction in size of wound | From Day 0 to week 4
  % change in surface area of wound; traced on OpSite Flexigrid ® film

SECONDARY OUTCOMES:
Presence of elevated protease activity in foot wound | Day 0
  Binary Yes/No; WOUNDCHEK™ Protease Status
Presence of elevated protease activity in foot wound | Day 14
  Binary Yes/No; WOUNDCHEK™ Protease Status
Presence of elevated protease activity in foot wound | Day 28
  Binary Yes/No; WOUNDCHEK™ Protease Status
Presence of bacterial protease activity in foot wound | Day 0, 14 and 28
  Binary Yes/No; WOUNDCHEK™ Bacterial Status
Presence of bacterial protease activity in foot wound | Day 14
  Binary Yes/No; WOUNDCHEK™ Bacterial Status
Presence of bacterial protease activity in foot wound | Day 28
  Binary Yes/No; WOUNDCHEK™ Bacterial Status
Clinical exam of wound | Day 0
  Classification as either infection or colonization according to Infectious Diseases Society of America classification
Presence of pathogenic bacteria in wound | Day 0
  Wound swabs cultured and bacteria identified
Presence of pathogenic bacteria in wound | Day 14
  Wound swabs cultured and bacteria identified
Presence of pathogenic bacteria in wound | Day 28
  Wound swabs cultured and bacteria identified
Reduction in size of wound | From Day 0 to Week 2
  % change in surface area of wound; traced on OpSite Flexigrid ® film

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Lavigne, Principal Investigator — CHU Nimes
Locations (4):
- France (4):
  - CH d'Alès, Alès
  - CH de Bagnols sur Céze, Bagnols-sur-Cèze
  - CHU de Montpellier, Montpellier
  - CHU de Nimes, Nîmes

IPD SHARING:
Plan to Share IPD: No